CLINICAL TRIAL: NCT05825781
Title: Randomized Double Blind Comparative Clinical Study Evaluating Pharmacokinetics and Safety in Single Intravenous Use of Pertuzumab (Manufactured by Mabscale, LLC) Compared to Perjeta® in Healthy Men
Brief Title: Study, Evaluating Pharmacokinetics, Immunogenicity and Safety Profiles of Pertuzumab Compared to Perjeta® in Healthy Man
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mabscale, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PERT-1/12102020
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Healthy Men
MeSH Terms: interventions — pertuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pertuzumab (manufactured by Mabscale, LLC) (Experimental): Eligible subjects (57 healthy men) will receive once Pertuzumab 420 mg/14 ml in 250 ml 0,9 % NaCl intravenous on the Visit 2. The following visits are the visits of safety and pharmacokinetics visits.
  Interventions: Drug: Pertuzumab
- Perjeta® (Active Comparator): Eligible subjects (57 healthy men) will receive once Perjeta® 420 mg/14 ml in 250 ml 0,9% NaCl intravenous on the Visit 2. The following visits are the visits of safety and pharmacokinetics visits.
  Interventions: Drug: Perjeta®

INTERVENTIONS:
Drug: Pertuzumab — i.v.
  Arms: Pertuzumab (manufactured by Mabscale, LLC)
Drug: Perjeta® — i.v.
  Arms: Perjeta®

SUMMARY:
PERT-1/12102020 is a double-blind randomized single-center clinical trial comparing pharmacokinetics, immunogenicity and safety profiles of Pertuzumab (manufactured by Mabscale, LLC) compared to Perjeta® in healthy men. The purpose of the study is to demonstrate equivalence of pharmacokinetics, immunogenicity and safety of Pertuzumab (manufactured by Mabscale, LLC) to Perjeta®.

DETAILED DESCRIPTION:
Pertuzumab is a recombinant humanized monoclonal antibody currently being developed by Mabscale LLC, as a proposed biosimilar to Perjeta®, which is approved as treatment in patients with metastatic breast cancer in combination with trastuzumab and docetaxel and in patients with non-metastatic breast cancer in combination with trastuzumab and chemotherapy. This randomized equivalence study is designed to meet the regulatory requirement for approval of a biosimilar product.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers, Men, 18 to 45 years old.
* Body mass index 18,5 - 30,0 kg/m2.
* Availability of written informed consent of the volunteer to participate in the study in accordance with applicable law.
* Volunteers should behave adequately, coherent speech should be observed.
* Volunteer consent to use an adequate method of contraception (barrier methods of contraception in combination with one of the following: non-hormonal intrauterine device; condom with intravaginal spermicide; cervical caps with spermicide; diaphragm with spermicide in the sexual partner) during the entire period of participation in the study and at least 6 months after the use of the study drug/comparator drug.
* The verified diagnosis is "healthy": the absence of pathology from the gastrointestinal tract, liver, kidneys, cardiovascular and bronchopulmonary systems, central nervous system (preliminary standard clinical, laboratory and instrumental studies did not reveal the presence of any diseases).
* Negative blood tests for HIV, syphilis and hepatitis (HBsAg and anti-HCV).
* LVEF ≥ 60% according to ECHO-CG.
* Negative urine test for drug and drug abuse.
* Negative breath alcohol test.

Exclusion Criteria:

1. Aggravated allergic anamnesis.
2. Hypersensitivity to pertuzumab and / or other substances that are part of the study drug.
3. Any vaccination up to 30 days before the expected date of administration of the drug according to medical history.
4. Drug intolerance.
5. Known intolerance to monoclonal antibody drugs (mouse, chimeric, humanized, human) according to medical history.
6. The results of laboratory analyzes provided for by the protocol are outside the established normative indicators of the investigator site.
7. Oncological diseases according to medical history.
8. Acute and chronic diseases of the cardiovascular, bronchopulmonary, neuroendocrine systems, as well as diseases of the gastrointestinal tract, liver, kidneys, hematopoietic, immune systems, mental illness.
9. More than 4 episodes of respiratory infections in the last 6 months prior to screening.
10. Surgical interventions on the gastrointestinal tract (with the exception of appendectomy).
11. Acute infectious diseases less than 4 weeks prior to study entry.
12. Taking drugs that have a pronounced effect on hemodynamics, liver function, etc. (barbiturates, omeprazole, cimetidine, etc.) less than 2 months before the start of this study.
13. Regular drug intake less than 2 weeks before the start of the study.
14. Systolic blood pressure less than 100 mm Hg. Art. or above 130 mm Hg. Art.; diastolic blood pressure less than 60 mm Hg. Art. or above 90 mm Hg. Art.; Heart rate less than 60 bpm or more than 90 bpm; respiratory rate less than 12 and more than 20 per minute
15. Donation of blood (450 ml of blood or more) less than 3 months before the start of the study.
16. Participation in clinical drug trials less than 3 months before the start of this study.
17. Taking more than 10 units of alcohol per week (where each unit is equal to 50 ml of strong alcoholic beverages or 500 ml of beer) or anamnestic information about alcoholism, drug addiction, drug abuse.
18. Smoking more than 10 cigarettes a day.
19. Any reason that, in the opinion of the investigator, would prevent a volunteer from participating in the study.
20. Mental, physical and other reasons that do not allow the subject adequately assess his behavior and correctly fulfill the conditions of the research protocol.
21. Special diet (eg vegetarian, vegan) or lifestyle (including night work and extreme physical activity such as heavy lifting) that may interfere with the study.
22. Volunteers who are expected to have problems with placing venous catheters or performing veinpuncture.
23. Depression according to medical history.
24. Insomnia according to medical history.
25. Inability to follow the schedule of study visits by a volunteer.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Concentration of pertuzumab in serum of subjects | Baseline up to 100 days after study drug administration

SECONDARY OUTCOMES:
Rate of subjects with antibodies against pertuzumab in serum | Baseline up to 100 days after study drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- Central Clinical Hospital "RZD-Medicina", Moscow, Russia

IPD SHARING:
Plan to Share IPD: No